CLINICAL TRIAL: NCT03754621
Title: What is the Rational Upper Limit for TSH and T4 During First and Second Trimester Pregnancy in West Black Sea Region of Turkey
Brief Title: Upper Limit for TSH of First and Second Trimester Pregnancy in Turkey
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bartin State Hospital (Other Government)
Responsible Party: Principal Investigator, Murat Yassa, Principal Investigator, Bartin State Hospital
Other Study IDs: IlSaglik2018-2
Record Dates: First submitted 2018-11-23; First posted 2018-11-27 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Thyroid; Thyroid Dysfunction; Hypothyroidism; Pregnancy Early
Keywords: TSH
MeSH Terms: conditions — Thyroid Diseases; Hypothyroidism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnants: 400 pregnant women with a singleton pregnancy, free of pre-existing thyroid disease, that do not use thyroid interfering medication, that did not undergo IVF treatment and are TPOAb negative. Serum thyroid functions tests will be obtained on the first visit.
  Interventions: Diagnostic Test: Serum thyroid functions tests

INTERVENTIONS:
Diagnostic Test: Serum thyroid functions tests — Serum TSH, fT3, fT4 and anti-TPO

SUMMARY:
Physiological changes necessitate the use of pregnancy-specific reference ranges for TSH and FT4 to diagnose thyroid dysfunction during pregnancy. Although many centers use fixed upper limits for TSH of 2.5 or 3.0 mU/L, this may lead to overdiagnosis or even overtreatment.

The new guidelines of the American Thyroid Association have considerably changed recommendations regarding thyroid function reference ranges in pregnancy accordingly. Any hospital or physician that is still using the 2.5 or 3.0 mU/l cut-off for TSH during pregnancy should evaluate their own lab-specific cut-offs.

The investigator's objective is to establish a rational reference range of serum TSH for diagnosis of subclinical hypothyroidism in the first and second trimester of pregnant women in west Black Sea region in Turkey.

DETAILED DESCRIPTION:
Serum thyroid function tests (including T3, T4, TSH, Anti-TPO) will be obtained from the singleton pregnancies in first and second trimester to determine the local specific normal ranges.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Free of pre-existing thyroid disease
* That do not use thyroid interfering medication
* That did not undergo IVF treatment
* TPOAb negative

Exclusion Criteria:

* Adolescent pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Turkish pregnant women living in Bartin Region of Turkey
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2018-10-15 (Actual); Primary Completion 2019-07-02 (Estimated); Study Completion 2019-07-15 (Estimated)

PRIMARY OUTCOMES:
TSH | Day 1
  Serum TSH (mU/I)

CONTACTS AND LOCATIONS:
Overall Officials: Murat Yassa, MD, Principal Investigator — Bartin State Hospital
Locations (1):
- Bartin State Hospital, Bartın, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Korevaar TIM. The upper limit for TSH during pregnancy: why we should stop using fixed limits of 2.5 or 3.0 mU/l. Thyroid Res. 2018 May 21;11:5. doi: 10.1186/s13044-018-0048-7. eCollection 2018. PMID 29942352